CLINICAL TRIAL: NCT01405963
Title: Randomized, Double-Blind, Placebo-Controlled, Parallel Design, Multiple-Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of AMG 157 in Subjects With Mild Atopic Asthma
Brief Title: Double-blind, Multiple Dose Study of Tezepelumab (AMG 157) in Adults With Mild Atopic Asthma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20101183
Record Dates: First submitted 2011-07-21; First posted 2011-07-29 (Estimated); Results first posted 2022-10-17 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2022-03

CONDITIONS: Asthma
Keywords: Amgen; AMG 157; Asthma
MeSH Terms: conditions — Asthma | interventions — tezepelumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Participants received placebo to tezepelumab administered by intravenous infusion on study days 1, 29, and 57.
  Interventions: Drug: Placebo
- Tezepelumab 700 mg (Experimental): Participants received 700 mg tezepelumab administered by intravenous infusion on study days 1, 29, and 57.
  Interventions: Biological: Tezepelumab

INTERVENTIONS:
Drug: Placebo — Administered in a 1-hour intravenous infusion
  Arms: Placebo
Biological: Tezepelumab — Administered in a 1-hour intravenous infusion
  Other Names: AMG 157; Tezspire
  Arms: Tezepelumab 700 mg

SUMMARY:
The purpose of this study is to assess the late and early asthmatic response after an allergen inhalation challenge in adults with mild atopic asthma after receiving multiple doses of tezepelumab (AMG 157), as well as the safety, tolerability, immunogenicity, and pharmacokinetics of multiple doses of tezepelumab in adults with mild atopic asthma.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects with history of mild atopic asthma between 18 and 60 years-of-age
* Body mass index (BMI) between 18 and 35 kg/m^2
* Normal or clinically acceptable physical examination (PE), clinical laboratory values, and electrocardiogram (ECG); clinically acceptable PE includes history of mild atopic asthma
* Used only inhaled short-acting β2-agonists infrequently to treat asthma
* No current exposure to allergens to which subject experiences asthmatic responses
* No other lung disease, exacerbations of asthma or lower respiratory tract infections for at least 6 weeks prior to screening
* Positive skin prick test to common aeroallergens at screening
* Additional inclusion criteria apply

Exclusion Criteria:

* History or evidence of a clinically significant disorder (including psychiatric), condition or disease that would pose a risk to subject safety or interfere with the study evaluation, procedures or completion;
* History or current medical conditions that are contraindicated for methacholine challenge, such as myocardial infarction or stroke within previous 3 months, known cardiac disease, uncontrolled hypertension and aortic or cerebral aneurysm
* Evidence of active or suspected bacterial, viral, fungal or parasitic infections within past 6 weeks
* Subject has know type I/II diabetes
* History of residential exposure to tuberculosis or has a positive purified protein derivative (PPD) or QuantiFERON test within 4 weeks before randomization
* Subject who has history of malignancy of any type within 5 years prior to enrollment
* Subjects tested positive for drugs/alcohol or nicotine use at screening
* Subjects tested positive for human immunodeficiency virus (HIV), hepatitis B or hepatitis C
* Additional exclusion criteria apply

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2011-10-31 (Actual); Primary Completion 2013-04-05 (Actual); Study Completion 2013-04-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (5):
- Canada (5):
  - Research Site, Calgary, Alberta
  - Research Site, Vancouver, British Columbia
  - Research Site, Hamilton, Ontario
  - Research Site, Sainte-Foy, Quebec
  - Research Site, Saskatoon, Saskatchewan

REFERENCES:
- [Derived] Gauvreau GM, O'Byrne PM, Boulet LP, Wang Y, Cockcroft D, Bigler J, FitzGerald JM, Boedigheimer M, Davis BE, Dias C, Gorski KS, Smith L, Bautista E, Comeau MR, Leigh R, Parnes JR. Effects of an anti-TSLP antibody on allergen-induced asthmatic responses. N Engl J Med. 2014 May 29;370(22):2102-10. doi: 10.1056/NEJMoa1402895. Epub 2014 May 20. PMID 24846652
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This proof-of-concept, randomized, double-blind, placebo-controlled study was conducted at 5 centers in Canada.
Pre-assignment Details: Participants were randomly assigned in a 1:1 ratio to receive tezepelumab or placebo.
Groups:
- Placebo: Participants received placebo administered by intravenous infusion on study days 1, 29, and 57.
Period: Overall Study
Arm/Group | Placebo | Tezepelumab 700 mg
Started | 15 | 16
Completed | 13 | 14
Not Completed | 2 | 2
Not completed — Moved Away | 2 | 0
Not completed — Adverse Event | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: Participants who received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Tezepelumab 700 mg | Total
Number analyzed (Participants) | 15 | 16 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.5 (11.2) | 30.8 (10.9) | 31.1 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 21
  Male | 4 | 6 | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Black or African American | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  White | 13 | 14 | 27
  Other | 1 | 0 | 1
Forced Expiratory Volume in 1 Second (FEV1) [Mean (Standard Deviation); unit: liters] | 3.335 (0.753) | 3.358 (0.865) | 3.346 (0.799)

OUTCOME MEASURES:

1. Primary Outcome: Maximum Percentage Decrease in Forced Expiratory Volume in 1 Second (FEV1) at 3 to 7 Hours Post Allergen Challenge
Description: Participants underwent allergen inhalation challenge on study days 42 and 84 to induce airway bronchoconstriction (measured by a fall in FEV1). FEV1 was measured prior to the challenge and between 3 to 7 hours post allergen challenge to assess late asthmatic response (LAR).
  The percent change in FEV1 from pre-challenge was calculated to each time point between 3 to 7 hours post challenge. The maximum percent decrease in FEV1 from pre-allergen challenge is the percent change in FEV1 representing the largest percentage decrease (or minimum percentage increase) from pre-allergen challenge FEV1 during late (3-7 hour) asthmatic response time frame.
Time Frame: Days 42 and 84 at pre-allergen challenge and at 180, 240, 300, 360, and 420 minutes (3-7 hours) post allergen challenge
Population: Participants who received at least 1 dose of study drug with available data on each day.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Tezepelumab 700 mg
Number analyzed (Participants) | 15 | 15
percent change
  Day 42 | -20.645 (11.554) | -16.949 (14.209)
  Day 84: number analyzed (Participants) | 12 | 14
  Day 84 | -19.366 (14.686) | -12.064 (9.131)
Statistical Analysis 1: Comparison: Placebo vs Tezepelumab 700 mg; Treatment difference in late asthmatic response at day 42 was evaluated using a repeated-measures analysis of covariance (ANCOVA) that included study treatment and study visit as independent variables, treatment by study visit as an interaction term, and the corresponding baseline value (as measured 14 days before the first dose of a study drug) as a model covariate; Test type: Other; p = 0.09, ANCOVA; Model includes treatment, visit, treatment by visit interaction as fixed effects and Day -14 value as covariate; Treatment Difference = 7.65, 95% CI 2-sided [-1.30 to 16.60] — Treatment difference estimate (tezepelumab minus placebo) is mean estimate based on ANCOVA
Statistical Analysis 2: Comparison: Placebo vs Tezepelumab 700 mg; Treatment difference in late asthmatic response at day 84 was evaluated using a repeated-measures ANCOVA that included study treatment and study visit as independent variables, treatment by study visit as an interaction term, and the corresponding baseline value (as measured 14 days before the first dose of a study drug) as a model covariate; Test type: Other; p = 0.02, ANCOVA; Model includes treatment, visit, treatment by visit interaction as fixed effects and Day -14 value as covariate; Treatment Difference = 9.91, 95% CI 2-sided [1.59 to 18.23] — Treatment difference estimate (tezepelumab minus placebo) is mean estimate based on ANCOVA

2. Primary Outcome: Time-Adjusted Area Under the Curve for the Percent Decrease From Pre-Allergen Challenge in Forced Expiratory Volume in 1 Second (FEV1) From 3 to 7 Hours Post Allergen Challenge
Description: Participants underwent allergen inhalation challenge on study days 42 and 84 to induce airway bronchoconstriction. FEV1 was measured prior to the challenge and between 3 to 7 hours post challenge to assess late asthmatic response (LAR).
  The percent change in FEV1 from pre-challenge was calculated to each time point between 3 to 7 hours post challenge. The area under the curve for the percent change at each time point was calculated using the linear trapezoidal rule, then time adjusted by dividing by the length of time over which the AUC was calculated.
Time Frame: Days 42 and 84 at pre-challenge and at 180, 240, 300, 360, and 420 minutes (3-7 hours) post challenge
Population: Participants who received at least 1 dose of study drug and with available AUC data on each day.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Tezepelumab 700 mg
Number analyzed (Participants) | 15 | 15
percent change
  Day 42 | 12.062 (8.231) | 9.321 (10.787)
  Day 84: number analyzed (Participants) | 12 | 14
  Day 84 | 11.864 (9.482) | 7.569 (7.069)
Statistical Analysis 1: Comparison: Placebo vs Tezepelumab 700 mg; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.11, ANCOVA; Model includes treatment, visit, treatment by visit interaction as fixed effects and day -14 value as covariate; Treatment Difference = -4.35, 95% CI 2-sided [-9.80 to 1.10] — Treatment difference estimate (tezepelumab minus placebo) is mean estimate based on ANCOVA
Statistical Analysis 2: Comparison: Placebo vs Tezepelumab 700 mg; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.07, ANCOVA; Model includes treatment, visit, treatment by visit interaction as fixed effects and day -14 value as covariate; Treatment Difference = -4.66, 95% CI 2-sided [-9.71 to 0.39] — Treatment difference estimate (tezepelumab minus placebo) is mean estimate based on ANCOVA

3. Secondary Outcome: Number of Participants With Adverse Events
Description: A serious adverse event is defined as an adverse event that meets at least 1 of the following serious criteria:
  * fatal,
  * life-threatening,
  * requires in-patient hospitalization or prolongation of existing hospitalization,
  * results in persistent or significant disability/incapacity,
  * congenital anomaly/birth defect, and/or
  * other medically important serious event. The severity of each adverse event was graded by the Investigator as mild, moderate, severe, life-threatening, or fatal according to the Common Terminology Criteria for Adverse Events (Version 4).
Time Frame: Up to 169 days
Population: Participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tezepelumab 700 mg
Number analyzed (Participants) | 15 | 16
Participants
  Any adverse event | 12 | 15
  Serious adverse event | 0 | 0
  Leading to discontinuation of study drug | 0 | 2
  Leading to discontinuation from study | 0 | 1
  Severe adverse events | 1 | 0
  Life-threatening adverse events | 0 | 0
  Fatal adverse events | 0 | 0
  Treatment-related adverse events | 3 | 4

4. Secondary Outcome: Number of Participants With Grade ≥ 3 Laboratory Values
Description: Laboratory toxicities were graded according to the Common Terminology Criteria for Adverse Events (Version 4) on a scale from grade 1 (mild) to 5 (death).
Time Frame: Up to 169 days
Population: Participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tezepelumab 700 mg
Number analyzed (Participants) | 15 | 16
Participants
  Any Grade ≥ 3 Laboratory Toxicity | 2 | 2
  Increased creatine kinase | 2 | 1
  Decreased lymphocytes | 0 | 1

5. Secondary Outcome: Number of Participants Who Developed Anti-tezepelumab Antibodies After Initiation of Treatment
Description: All study samples (tezepelumab and placebo) were tested using an electrochemiluminescence (ECL) based immunoassay to detect and confirm the presence of antibodies capable of binding to tezepelumab. Samples identified as positive in the immunoassay were tested in a receptor-binding ECL-based assay to detect neutralizing or inhibitory effects toward tezepelumab.
  The number of participants with positive anti-tezepelumab binding antibodies / neutralizing antibodies at any time post-baseline with a negative or no result at baseline is reported.
Time Frame: Days 29, 57, 85, 113, and 169
Population: Participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tezepelumab 700 mg
Number analyzed (Participants) | 15 | 16
Participants
  Anti-tezepelumab binding antibodies | 1 | 0
  Anti-tezepelumab neutralizing antibodies | 0 | 0

6. Secondary Outcome: Maximum Percentage Decrease in FEV1 From 0 to 2 Hours Post Allergen Challenge
Description: Participants underwent allergen inhalation challenge on study days 42 and 84 to induce airway bronchoconstriction. FEV1 was measured prior to the challenge and between 0 to 2 hours post challenge to assess early asthmatic response (EAR).
  The maximum percent decrease in FEV1 from pre-allergen challenge is the percent change in FEV1 representing the largest percentage decrease (or minimum percentage increase) from pre-allergen challenge FEV1 during early (0-2 hour) asthmatic response time frame.
Time Frame: Days 42 and 84 at pre-allergen challenge and at 10, 20, 30, 45, 60, 90, and 120 minutes (0-2 hours) post allergen challenge
Population: Participants who received at least 1 dose of study drug with available data on each day.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Tezepelumab 700 mg
Number analyzed (Participants) | 15 | 15
percent change
  Day 42 | -33.296 (10.084) | -22.501 (15.001)
  Day 84: number analyzed (Participants) | 13 | 14
  Day 84 | -33.160 (15.280) | -20.990 (13.393)
Statistical Analysis 1: Comparison: Placebo vs Tezepelumab 700 mg; Treatment difference in early asthmatic response at day 42 was evaluated using a repeated-measures ANCOVA that included study treatment and study visit as independent variables, treatment by study visit as an interaction term, and the corresponding baseline value (as measured 14 days before the first dose of a study drug) as a model covariate; Test type: Other; p = 0.05, ANCOVA; Model includes treatment, visit, treatment by visit interaction as fixed effects and Day -14 value as covariate; Treatment Difference = 8.57, 95% CI 2-sided [0.01 to 17.13] — Treatment difference estimate (tezepelumab minus placebo) is mean estimate based on ANCOVA
Statistical Analysis 2: Comparison: Placebo vs Tezepelumab 700 mg; Treatment difference in early asthmatic response at day 84 was evaluated using a repeated-measures ANCOVA that included study treatment and study visit as independent variables, treatment by study visit as an interaction term, and the corresponding baseline value (as measured 14 days before the first dose of a study drug) as a model covariate; Test type: Other; p = 0.06, ANCOVA; Model includes treatment, visit, treatment by visit interaction as fixed effects and Day -14 value as covariate; Treatment Difference = 10.27, 95% CI 2-sided [-0.46 to 21.00] — Treatment difference estimate (tezepelumab minus placebo) is mean estimate based on ANCOVA

7. Secondary Outcome: Time-Adjusted AUC for the Percent Decrease From Pre-Allergen Challenge in FEV1 From 0 to 2 Hours Post Allergen Challenge
Description: Participants underwent allergen inhalation challenge on study days 42 and 84 to induce airway bronchoconstriction. FEV1 was measured prior to the challenge and between 0 to 2 hours post challenge to assess early asthmatic response (EAR).
  The percent change in FEV1 from pre-allergen challenge was calculated to each time point between 0 to 2 hours post challenge. The area under the curve for the percent change at each time point was calculated using the linear trapezoidal rule, then time adjusted by dividing by the length of time over which the AUC was calculated.
Time Frame: Days 42 and 84 at pre-challenge and at 10, 20, 30, 45, 60, 90, and 120 minutes (0-2 hours) post challenge
Population: Participants who received at least 1 dose of study drug and with available AUC data on each day.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Tezepelumab 700 mg
Number analyzed (Participants) | 15 | 15
percent change
  Day 42 | 18.592 (8.432) | 11.284 (11.509)
  Day 84: number analyzed (Participants) | 13 | 14
  Day 84 | 20.179 (10.973) | 11.297 (10.708)
Statistical Analysis 1: Comparison: Placebo vs Tezepelumab 700 mg; [analysis description as in outcome 6, analysis 1]; Test type: Other; p = 0.03, ANCOVA; Model includes treatment, visit, treatment by visit interaction as fixed effects and day -14 value as covariate; Treatment Difference = -6.08, 95% CI 2-sided [-11.56 to -0.60] — Treatment difference estimate (tezepelumab minus placebo) is mean estimate based on ANCOVA
Statistical Analysis 2: Comparison: Placebo vs Tezepelumab 700 mg; [analysis description as in outcome 6, analysis 2]; Test type: Other; p = 0.03, ANCOVA; Model includes treatment, visit, treatment by visit interaction as fixed effects and day -14 value as covariate; Treatment Difference = -7.44, 95% CI 2-sided [-14.22 to -0.66] — Treatment difference estimate (tezepelumab minus placebo) is mean estimate based on ANCOVA

8. Secondary Outcome: Minimum FEV1 From 0 to 2 Hours Post Allergen Challenge
Description: Participants underwent allergen inhalation challenge on study days 42 and 84 to induce airway bronchoconstriction. FEV1 was measured prior to the challenge and between 0 to 2 hours post challenge to assess early asthmatic response (EAR).
  The minimum FEV1 post onset of the allergen challenge for EAR is defined as the smallest value of FEV1 measured during 0 to 2 hours post allergen challenge.
Time Frame: Days 42 and 84 at 10, 20, 30, 45, 60, 90, and 120 minutes (0-2 hours) post allergen challenge
Population: Participants who received at least 1 dose of study drug with available data on each day.
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Placebo | Tezepelumab 700 mg
Number analyzed (Participants) | 15 | 15
liters
  Day 42 | 2.211 (0.589) | 2.682 (0.839)
  Day 84: number analyzed (Participants) | 13 | 14
  Day 84 | 2.184 (0.720) | 2.774 (0.826)
Statistical Analysis 1: Comparison: Placebo vs Tezepelumab 700 mg; [analysis description as in outcome 6, analysis 1]; Test type: Other; p = 0.05, ANCOVA; Model includes treatment, visit, treatment by visit interaction as fixed effects and Day -14 value as covariate; Treatment Difference = 0.33, 95% CI 2-sided [-0.01 to 0.68] — Treatment difference estimate (tezepelumab minus placebo) is mean estimate based on ANCOVA
Statistical Analysis 2: Comparison: Placebo vs Tezepelumab 700 mg; [analysis description as in outcome 6, analysis 2]; Test type: Other; p = 0.08, ANCOVA; Model includes treatment, visit, treatment by visit interaction as fixed effects and Day -14 value as covariate; Treatment Difference = 0.39, 95% CI 2-sided [-0.06 to 0.84] — Treatment difference estimate (tezepelumab minus placebo) is mean estimate based on ANCOVA

9. Secondary Outcome: Time-Adjusted AUC for FEV1 From 0 to 2 Hours Post Allergen Challenge
Description: Participants underwent allergen inhalation challenge on study days 42 and 84 to induce airway bronchoconstriction. FEV1 was measured prior to the challenge and between 0 to 2 hours post challenge to assess early asthmatic response (EAR).
  The area under the curve for the FEV1 between 0 to 2 hours post allergen challenge was calculated using the linear trapezoidal rule, then time adjusted by dividing by the length of time over which the AUC was calculated.
Time Frame: Days 42 and 84 at pre-challenge and at 10, 20, 30, 45, 60, 90, and 120 minutes (0-2 hours) post challenge
Population: Participants who received at least 1 dose of study drug and with available AUC data on each day.
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Placebo | Tezepelumab 700 mg
Number analyzed (Participants) | 15 | 15
liters
  Day 42 | 2.709 (0.695) | 3.076 (0.844)
  Day 84: number analyzed (Participants) | 13 | 14
  Day 84 | 2.607 (0.681) | 3.120 (0.856)
Statistical Analysis 1: Comparison: Placebo vs Tezepelumab 700 mg; [analysis description as in outcome 6, analysis 1]; Test type: Other; p = 0.03, ANCOVA; Model includes treatment, visit, treatment by visit interaction as fixed effects and day -14 value as covariate; Treatment Difference = 0.28, 95% CI 2-sided [0.03 to 0.53] — Treatment difference estimate (tezepelumab minus placebo) is mean estimate based on ANCOVA
Statistical Analysis 2: Comparison: Placebo vs Tezepelumab 700 mg; [analysis description as in outcome 6, analysis 2]; Test type: Other; p = 0.06, ANCOVA; Model includes treatment, visit, treatment by visit interaction as fixed effects and day -14 value as covariate; Treatment Difference = 0.33, 95% CI 2-sided [-0.01 to 0.66] — Treatment difference estimate (tezepelumab minus placebo) is mean estimate based on ANCOVA

10. Secondary Outcome: Minimum FEV1 From 3 to 7 Hours Post Allergen Challenge
Description: Participants underwent allergen inhalation challenge on study days 42 and 84 to induce airway bronchoconstriction. FEV1 was measured prior to the challenge and between 3 to 7 hours post challenge to assess late asthmatic response (LAR).
  The minimum FEV1 post allergen challenge for LAR is defined as the smallest value of FEV1 measured during 3 to 7 hours post allergen challenge.
Time Frame: Days 42 and 84 at 180, 240, 300, 360, and 420 minutes (3-7 hours) post allergen challenge
Population: Participants who received at least 1 dose of study drug with available data on each day.
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Placebo | Tezepelumab 700 mg
Number analyzed (Participants) | 15 | 15
liters
  Day 42 | 2.659 (0.778) | 2.943 (1.036)
  Day 84: number analyzed (Participants) | 12 | 14
  Day 84 | 2.627 (0.864) | 3.097 (0.827)
Statistical Analysis 1: Comparison: Placebo vs Tezepelumab 700 mg; Treatment difference in late asthmatic response at day 42 was evaluated using a repeated-measures ANCOVA that included study treatment and study visit as independent variables, treatment by study visit as an interaction term, and the corresponding baseline value (as measured 14 days before the first dose of a study drug) as a model covariate; Test type: Other; p = 0.01, ANCOVA; Model includes treatment, visit, treatment by visit interaction as fixed effects and Day -14 value as covariate; Treatment Difference = 0.41, 95% CI 2-sided [0.12 to 0.70] — Treatment difference estimate (tezepelumab minus placebo) is mean estimate based on ANCOVA
Statistical Analysis 2: Comparison: Placebo vs Tezepelumab 700 mg; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.01, ANCOVA; Model includes treatment, visit, treatment by visit interaction as fixed effects and Day -14 value as covariate; Treatment Difference = 0.42, 95% CI 2-sided [0.11 to 0.72] — Treatment difference estimate (tezepelumab minus placebo) is mean estimate based on ANCOVA

11. Secondary Outcome: Time-Adjusted AUC for FEV1 From 3 to 7 Hours Post Allergen Challenge
Description: Participants underwent allergen inhalation challenge on study days 42 and 84 to induce airway bronchoconstriction. FEV1 was measured prior to the challenge and between 3 to 7 hours post allergen challenge to assess late asthmatic response (LAR).
  The area under the curve for the FEV1 between 3 to 7 hours post allergen challenge was calculated using the linear trapezoidal rule, then time adjusted by dividing by the length of time over which the AUC was calculated.
Time Frame: Days 42 and 84 at pre-challenge and at 180, 240, 300, 360, and 420 minutes (3-7 hours) post challenge.
Population: Participants who received at least 1 dose of study drug and with available AUC data on each day.
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Placebo | Tezepelumab 700 mg
Number analyzed (Participants) | 15 | 15
liters
  Day 42 | 2.940 (0.781) | 3.188 (0.994)
  Day 84: number analyzed (Participants) | 12 | 14
  Day 84 | 2.853 (0.780) | 3.252 (0.831)
Statistical Analysis 1: Comparison: Placebo vs Tezepelumab 700 mg; [analysis description as in outcome 10, analysis 1]; Test type: Other; p = 0.02, ANCOVA; Model includes treatment, visit, treatment by visit interaction as fixed effects and day -14 value as covariate; Treatment Difference = 0.24, 95% CI 2-sided [0.04 to 0.45] — Treatment difference estimate (tezepelumab minus placebo) is mean estimate based on ANCOVA
Statistical Analysis 2: Comparison: Placebo vs Tezepelumab 700 mg; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.15, ANCOVA; Model includes treatment, visit, treatment by visit interaction as fixed effects and day -14 value as covariate; Treatment Difference = 0.18, 95% CI 2-sided [-0.07 to 0.44] — Treatment difference estimate (tezepelumab minus placebo) is mean estimate based on ANCOVA

12. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) of Tezepelumab
Description: The PK parameter Cmax was estimated based on the serum concentrations of tezepelumab using noncompartmental methods. The concentration of tezepelumab in human serum was measured using a validated ELISA. The lower limit of quantification of the assay was 10 ng/mL.
Time Frame: First dose: Day 1 at predose and 1 and 4 hours postdose, and days 4, 8, 15, and 29 (predose); Last dose: Day 57 predose, 1 and 4 hours postdose, and at days 60, 64, 71, 83, 84, 85, 113, and 169.
Population: The pharmacokinetic (PK) parameter analysis set includes participants for whom pharmacokinetic parameter estimates could be derived after first dose and after last dose.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Tezepelumab 700 mg
Number analyzed (Participants) | 16
μg/mL
  First dose | 262 (73)
  Last dose: number analyzed (Participants) | 14
  Last dose | 325 (81)

13. Secondary Outcome: Time of Maximum Observed Concentration (Tmax) of Tezepelumab
Description: The PK parameter Tmax was estimated based on the serum concentrations of tezepelumab using noncompartmental methods. The concentration of tezepelumab in human serum was measured using a validated ELISA. The lower limit of quantification of the assay was 10 ng/mL.
Time Frame: as for outcome 12
Population: The PK parameter analysis set includes participants for whom pharmacokinetic parameter estimates could be derived after first dose and after last dose.
Measure: Median (Full Range); unit: hours
Arm/Group | Tezepelumab 700 mg
Number analyzed (Participants) | 16
hours
  First dose | 2.1 [1.0 to 5.2]
  Last dose: number analyzed (Participants) | 14
  Last dose | 2.0 [1.1 to 5.0]

14. Secondary Outcome: Minimum Observed Serum Concentration (Cmin) of Tezepelumab
Description: The PK parameter Cmin was estimated based on the serum concentrations of tezepelumab using noncompartmental methods. The concentration of tezepelumab in human serum was measured using a validated ELISA. The lower limit of quantification of the assay was 10 ng/mL.
Time Frame: as for outcome 12
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Tezepelumab 700 mg
Number analyzed (Participants) | 16
μg/mL
  First dose | 60.7 (20.8)
  Last dose: number analyzed (Participants) | 14
  Last dose | 17.7 (13.4)

15. Secondary Outcome: Area Under the Concentration-time Curve Over the Dosing Interval (AUCtau) for Tezepelumab
Description: The PK parameter AUCtau was estimated based on the serum concentrations of tezepelumab using noncompartmental methods.
  The dosing interval (tau) was 28 days. The concentration of tezepelumab in human serum was measured using a validated ELISA. The lower limit of quantification of the assay was 10 ng/mL.
Time Frame: First dose: Day 1 at predose and 1 and 4 hours postdose and days 4, 8, 15, and 29 (predose); Last dose: Day 57 predose, 1 and 4 hours postdose, and at days 60, 64, 71, 83, 84, and 85.
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: day*μg/mL
Arm/Group | Tezepelumab 700 mg
Number analyzed (Participants) | 16
day*μg/mL
  First dose | 2730 (700)
  Last dose: number analyzed (Participants) | 14
  Last dose | 4420 (1250)

16. Secondary Outcome: Accumulation Ratio Based on AUCtau
Description: Accumulation ratio (AR) based on AUCtau was calculated as AUCtau after last dose / AUCtau after first dose.
Time Frame: as for outcome 15
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Tezepelumab 700 mg
Number analyzed (Participants) | 14
ratio | 1.64 (0.25)

17. Secondary Outcome: Accumulation Ratio Based on Cmax
Description: Accumulation ratio based on Cmax calculated as Cmax after last dose / Cmax after first dose.
Time Frame: as for outcome 12
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Tezepelumab 700 mg
Number analyzed (Participants) | 14
ratio | 1.31 (0.25)

18. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero to Infinity (AUCinf) After Last Dose for Tezepelumab
Description: The PK parameter AUCinf was estimated based on the serum concentrations of tezepelumab using noncompartmental methods. The concentration of tezepelumab in human serum was measured using a validated ELISA. The lower limit of quantification of the assay was 10 ng/mL.
Time Frame: Day 57 predose, 1 and 4 hours postdose, and at days 60, 64, 71, 83, 84, 85, 113, and 169.
Population: The PK parameter analysis set includes participants for whom pharmacokinetic parameter estimates could be derived after last dose.
Measure: Mean (Standard Deviation); unit: day*μg/mL
Arm/Group | Tezepelumab 700 mg
Number analyzed (Participants) | 14
day*μg/mL | 8620 (2440)

19. Secondary Outcome: Terminal Half-life (t1/2z) of Tezepelumab After Last Dose
Description: The PK parameter t1/2,z was estimated based on the serum concentrations of tezepelumab using noncompartmental methods. The concentration of tezepelumab in human serum was measured using a validated ELISA. The lower limit of quantification of the assay was 10 ng/mL.
Time Frame: Day 57 predose, 1 and 4 hours postdose, and at days 60, 64, 71, 83, 84, 85, 113, and 169.
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Tezepelumab 700 mg
Number analyzed (Participants) | 14
days | 28.0 (4.2)

ADVERSE EVENTS:
Time Frame: 169 days
Arm/Group | Placebo | Tezepelumab 700 mg
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/16
Other Adverse Events (participants affected / at risk) | 12/15 | 15/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=15) | Tezepelumab 700 mg (N=16)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 1
Ear pain (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Eye pruritus (Eye disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 1 | 1
Influenza like illness (General disorders) | 1 | 0
Malaise (General disorders) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 1 | 0
Labyrinthitis (Infections and infestations) | 1 | 0
Laryngitis (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 2 | 0
Nasopharyngitis (Infections and infestations) | 4 | 4
Pharyngitis (Infections and infestations) | 1 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 1
Rhinitis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 1
Headache (Nervous system disorders) | 3 | 2
Hypoaesthesia (Nervous system disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.